CLINICAL TRIAL: NCT04270461
Title: A Phase I Clinical Trial of NKG2D-based CAR T-cells Injection for Subjects With Relapsed/Refractory NKG2DL+ Solid Tumors
Brief Title: NKG2D-based CAR T-cells Immunotherapy for Patient With r/r NKG2DL+ Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study is withdrawn because of administrative reasons
Sponsor: Jiujiang University Affiliated Hospital (Other Government)
Collaborators: KAEDI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JiujiangUH
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Hepatocellular Carcinoma; Glioblastoma; Medulloblastoma; Colon Cancer
Keywords: NKG2D-based CAR T-cells; solid tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular; Glioblastoma; Medulloblastoma; Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arms (Experimental): NKG2D-based CAR T-cells Injection; Dosage:1-10x10^6/kg, 70ml/time, The CAR-T cells will be administered by i.v. or hepatic portal artery injection over 20-30 minutes Frequency: total one time
  Interventions: Biological: NKG2D-based CAR T-cells

INTERVENTIONS:
Biological: NKG2D-based CAR T-cells — Autologous genetically modified anti-NKG2DLs CAR transduced T cells
  Other Names: KD-025 CAR T-cells

SUMMARY:
The primary objective of this study is to evaluate the safety and clinical activity of NKG2D-based CAR-T cells infusion in the treatment of relapsed/refractory NKG2DL+ solid tumors.

DETAILED DESCRIPTION:
The preclinical study clarified that NKG2D-based CAR-T cells showed strong cytotoxicity against NKG2DL+ cell lines in vitro as well as a therapeutic effect against NKG2DL+ cell xenografts in vivo. In addition, the data also demonstrated the safety of NKG2D-based CAR-T therapy. NKG2D-based CAR-T represent a potentially effective and safety therapeutic approach for patient with relapsed/refractory NKG2DL+ solid tumors. In this trial, the investigators researched the safety of administering NKG2D-based CAR-T which generated with CD8 hinge region and transmembrane region, 4-1BB costimulatory region and CD3 zeta region. The investigators also assessed that disease response was determined within the context of a phase I trial.

ELIGIBILITY:
Inclusion criteria:

1. Men or women≥18 years old,
2. Patient with NKG2DL+ cell tumors confirmed by pathology and histology，
3. Fail or unwilling to receive first-line treatment,
4. Disease must be measurable according to the corresponding guidelines,
5. Main organs function normally and meet following requirements:

   Routine blood index（No Blood transfusion within 14 days） 1)HB≥90g/L; 2)ANC≥1.5×109/L; 3)PLT≥75×109/L； Serum biochemicals index 1) BIL <1.5 upper normal limit (ULN); 2) ALT and AST<2.5×ULN; In the case of liver metastasis, ALT and AST<5×ULN; 3) Serum Cr≤1×ULN, endogenous creatinine clearance≥50ml/min (Cockcroft-Gault formula); 4) ECOG physical condition score: 0-2
6. Expected survival time ≥3 months,
7. Patient with adequate bone marrow reserve, hepatic and renal functions,
8. No other uncontrolled diseases such as lung, kidney and liver infection before enrollment,
9. Women of child-bearing age must undergo a negative pregnancy test (serum or urine) within 7 days prior to enrollment and voluntarily use appropriate methods of contraception during the observation period and within 8 weeks after the last dose; men should agree to contraception during the observation period and within 8 weeks of the last dose,
10. Patients voluntarily participated in this trial and sign the informed consent form,
11. Patients with compliance and expected to follow up the efficacy and adverse reactions as required by the protocol.

Exclusion criteria:

1. Pregnant or lactating women,
2. Patients who need to use systemic steroids at the same time,
3. Under following treatment conditions currently: 1) during the other anti- tumor clinical observation period within 14 days before blood collection; 2) patient has not recovered from acute side effects of the previous treatment;
4. Receive radiotherapy within 4 weeks before enrollment,
5. Patients who received any other cell therapy before,
6. Patients with unqualified T cell amplification efficiency,
7. Uncontrolled symptoms or other illnesses, including but not limited to infection, congestive heart failure, unstable angina, arrhythmia, psychosis,
8. Patients with severe acute allergic reactions,
9. Patients who have received other cell therapies,
10. Other serious conditions that may limit patient's participation in the study.

Detailed disease specific criteria exist and can be discussed with contacts listed below.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with severe cytokine release syndrome(CRS) as a Measure of Safety and Tolerability. | 0 to 28 days post infusion
  The severe CRS post KD-025 CAR-T cells treatment will be evaluated and the maximum tolerated dose will be determined.
Copies numbers of CAR | 1 year post infusion
  Copies numbers of CAR in peripheral blood (PB)

SECONDARY OUTCOMES:
overall survival (OS) | 2 years post infusion
  For all subjects, overall survival refers to the period from being included in the test group to death caused by any reason
Progress Free Survival (PFS) | 2 years post infusion
  Progress Free Survival after administration
Duration of response, (DoR) | 2 years post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Changchun Cai, Study Director — Affiliated hospital of jiujiang university
Locations (1):
- Affiliated hospital of jiujiang university, Jiujiang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No